CLINICAL TRIAL: NCT05450939
Title: Analysis of Hemodynamic Characteristics Using Signal Intensity Gradient of Brain Magnetic Resonance Imaging in Patients With Subarachnoid Hemorrhage After Rupture of Intracranial Aneurysm
Brief Title: Characteristics of Signal Intensity Gradient in Subarachnoid Hemorrhage After Aneurysmal Rupture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Chan-Hyuk Lee, Principal Investigator, Chonbuk National University Hospital
Other Study IDs: SIGSAH
Record Dates: First submitted 2022-06-29; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Aneurysmal Rupture
Keywords: Signal intensity gradient; Wall shear stress; Aneurysmal rupture; Time-of-Flight MRI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ruptured group: Group of subarachnoid hemorrhage after rupture of intracranial aneurysm
  Interventions: Diagnostic Test: Signal intensity gradient
- Unruptured group: Group of inexperience of aneurysmal rupture during specific period
  Interventions: Diagnostic Test: Signal intensity gradient

INTERVENTIONS:
Diagnostic Test: Signal intensity gradient — In time-of-flight (TOF) MRA, The signal intensities at the iso-point (Φa; signal intensity at position A [Xa] along the arterial contour line) and at the inner point (Φb; signal intensity at position B [Xb]) were calculated by using a trilinear interpolation algorithm based on the positions and signal intensities in the eight neighboring voxels. The signal intensities of TOF-MRA were normalized to eliminate the offset and scale effects across the MRA datasets of participants. For each iso-point (position A), the SIG was calculated from the difference in signal intensities between points A and B as follows:
  Scalar SIG, SI/mm = (Φb - Φa) / │Xb - Xa│ (1)
  Vector SIG, SI/mm = (Φb - Φa) n / │Xb - Xa│ (2)

SUMMARY:
10-20% of patients with subarachnoid hemorrhage die before they arrive at the hospital, and about 25% die within 24 hours. About 1% of patients are diagnosed with cerebral aneurysms in imaging tests for health checkups, and many of them experience aneurysmal rupture during their lifetime, so it is not a rare disease. Wall shear stress is known to be a factor that reflects the state of blood vessels, and particularly plays an important role in the patency of the intima of blood vessels. In the meantime, computed fluid dynamics (CFD), a representative method for calculating wall shear stress, assumes a virtual rigid pipe and applies a preset value. This does not accurately reflect the physiological and dynamic state of the actual blood vessel. The investigators intend to measure the patient's wall shear stress using the SIG of the MRA-TOF technique, which reflects the physiological characteristics of individual patients, and to analyze the association with rupture of the intracranial aneurysm.

ELIGIBILITY:
<Ruptured group>

Inclusion Criteria:

1) Patients over 18 years of age who visited our hospital for acute subarachnoid hemorrhage due to rupture of a intracranial aneurysm (2) Among patients satisfying (1), who had intracranial magnetic resonance imaging (time-of-flight (TOF) technique applied; diffusion-weighted imaging, including apparent diffusion coefficient) before subarachnoid hemorrhage occurred.

Exclusion Criteria:

1. Patients under the age of 18
2. Patients with subarachnoid hemorrhage due to causes other than rupture of intracranial aneurysm
3. Patients with poor imaging quality due to artifacts caused by patient movement during brain magnetic resonance imaging examination

<Unruptured group>

Inclusion Criteria:

1. Magnetic resonance imaging performed during the screening period (Time-of-Flight (TOF) technique is applied to intracranial vessel imaging; It also includes diffusion-weighted imaging and apparent diffusion coefficient)
2. Patients diagnosed with unruptured intracranial aneurysm in the final reading of brain MR test
3. Patients who remain without aneurysmal rupture on follow-up intracranial magnetic resonance imaging

Exclusion Criteria:

1. Patients under the age of 18
2. Patients with poor imaging quality due to artifacts caused by patient movement during brain magnetic resonance imaging examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visited health checkup program or neurology clinic (unruptured group), or emergency department (ruptured group) of a tertiary center
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-11-25 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Degree of signal intensity gradient in aneurysmal sac | Average 4-6 years
  The investigators will measure the degree of signal intensity gradient (SIG) from brain TOF-MRA in aneurysmal sac.
  The measured SIG in ruptured group would be lower than that in unruptured group.

CONTACTS AND LOCATIONS:
Overall Officials: Chan-Hyuk Lee, Dr., Principal Investigator — Jeonbuk National University Hospital
Locations (1):
- Jeonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han KS, Lee SH, Ryu HU, Park SH, Chung GH, Cho YI, Jeong SK. Direct Assessment of Wall Shear Stress by Signal Intensity Gradient from Time-of-Flight Magnetic Resonance Angiography. Biomed Res Int. 2017;2017:7087086. doi: 10.1155/2017/7087086. Epub 2017 Aug 16. PMID 28900625
- [Background] Suzuki T, Stapleton CJ, Koch MJ, Tanaka K, Fujimura S, Suzuki T, Yanagisawa T, Yamamoto M, Fujii Y, Murayama Y, Patel AB. Decreased wall shear stress at high-pressure areas predicts the rupture point in ruptured intracranial aneurysms. J Neurosurg. 2019 Mar 15;132(4):1116-1122. doi: 10.3171/2018.12.JNS182897. Print 2020 Apr 1. PMID 30875692
- [Background] Lee WJ, Jeong SK, Han KS, Lee SH, Ryu YJ, Sohn CH, Jung KH. Impact of Endothelial Shear Stress on the Bilateral Progression of Unilateral Moyamoya Disease. Stroke. 2020 Mar;51(3):775-783. doi: 10.1161/STROKEAHA.119.028117. Epub 2019 Dec 20. PMID 31856692
- [Derived] Lee CH, Kwak HS, Kang HS, Jung KH, Jeong SK. Geometric versus Hemodynamic Indexes for Rupture-Destined Aneurysms: A Retrospective Cohort and a Repeated-Measures Study. Cerebrovasc Dis. 2024;53(3):327-334. doi: 10.1159/000533167. Epub 2023 Sep 11. PMID 37696264